CLINICAL TRIAL: NCT06917950
Title: Effect of Roxadustat on Bone and Neuropsychiatric Aspects in End Stage Kidney Disease Patients on Hemodialysis
Brief Title: Roxadustat for Bone and Neuropsychiatric Aspects in Hemodialysis Patients
Acronym: ROXA-BN-HD
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mostafa Ibrahim Alsayed Alaskary, Principal Investigator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MD.24.08.877
Record Dates: First submitted 2025-03-27; First posted 2025-04-09 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Kidney Failure,Chronic; Anemia in End Stage Renal Disease; Depression Anxiety Disorder
Keywords: Roxadustat; Hemodialysis; Renal Anemia; Bone Mineral Density (BMD); Quantitative Computed Tomography (QCT); Neuropsychiatric; Musculoskeletal Ultrasound (MSK-US)
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — roxadustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Roxadustat Group (Experimental): Participants randomized to this arm will receive oral Roxadustat (Evernzo) three times per week according to standard dosing guidelines for managing anemia in hemodialysis patients. Participants will continue standard care for other conditions but will discontinue other erythropoiesis-stimulating agents (ESAs). Dosing may be adjusted based on hemoglobin response as per protocol and product labeling.
  Interventions: Drug: Roxadustat
- Conventional Treatment Group (Active Comparator): Participants randomized to this arm will continue receiving their conventional management for renal anemia, typically including erythropoiesis-stimulating agents (ESAs) and/or intravenous iron, as determined by standard clinical practice at the study site. Participants will receive standard care for all other conditions.
  Interventions: Drug: Conventional Anemia Management

INTERVENTIONS:
Drug: Roxadustat — Oral hypoxia-inducible factor prolyl hydroxylase inhibitor (HIF-PHI). Administered orally three times per week. Dosage will be initiated and adjusted according to prescribing guidelines for treating anemia associated with chronic kidney disease in patients on dialysis based on hemoglobin levels.
  Arms: Roxadustat Group
Drug: Conventional Anemia Management — Standard of care treatment for renal anemia, typically involving administration of erythropoiesis-stimulating agents (ESAs, e.g., epoetin, darbepoetin) and/or intravenous iron supplementation. Dosing and specific agents used are per standard clinical practice at the study site and adjusted based on hemoglobin levels and iron status according to prevailing guidelines.
  Arms: Conventional Treatment Group

SUMMARY:
People with severe kidney failure who need regular hemodialysis treatment often experience several health problems. These include anemia (low red blood cell count), issues with their bone health (sometimes called mineral and bone disease), and mental health challenges like depression and anxiety. They may also have problems with their nerves and muscles.

Roxadustat is a newer medicine, taken as a pill, used to treat anemia caused by kidney disease. It works differently than the standard injectable medications often used.

This study aims to investigate if Roxadustat has effects beyond treating anemia in hemodialysis patients. Specifically, researchers want to see if taking Roxadustat affects patients' bone health (measured by bone density scans and blood tests) and their psychological well-being (looking at symptoms of depression and anxiety using questionnaires). The study will also use ultrasound to look at potential changes in nerves and muscles.

The study will enroll 46 patients on hemodialysis. Patients will be randomly assigned (like flipping a coin) into two groups. One group (23 patients) will receive Roxadustat three times a week, while the other group (23 patients) will continue receiving their usual conventional treatment for anemia.

All patients will be followed for 6 months. During this time, they will have regular blood tests, bone density scans (using a technique called QCT), nerve and muscle ultrasound examinations, and will complete questionnaires about their mood.

Researchers will compare the results between the two groups to understand the effects of Roxadustat on bone, mood, anxiety, and neuromuscular aspects in patients undergoing hemodialysis

DETAILED DESCRIPTION:
Background:

Chronic kidney disease (CKD) is a major global health issue. Renal anemia is a frequent and significant complication, affecting over 90% of patients with end-stage kidney disease (ESKD) requiring hemodialysis. Anemia in this population contributes to reduced quality of life, increased cardiovascular events, hospitalizations, and mortality. While erythropoiesis-stimulating agents (ESAs) combined with iron supplementation are the standard first-line treatment, concerns exist regarding potential adverse events associated with high ESA doses and hyporesponsiveness in some patients, highlighting the need for alternative therapeutic strategies.

Roxadustat is an orally administered hypoxia-inducible factor prolyl hydroxylase inhibitor (HIF-PHI). By inhibiting HIF prolyl hydroxylase enzymes, Roxadustat mimics the body's response to hypoxia, leading to increased stabilization and activity of HIF. This, in turn, promotes endogenous erythropoietin (EPO) production, improves iron metabolism and mobilization, and effectively treats renal anemia.

Rationale:

Beyond anemia, ESKD patients face a high burden of other complications, including mineral and bone disorders (CKD-MBD) and neuropsychiatric issues such as depression, anxiety, and neuromuscular dysfunction. The HIF pathway, targeted by Roxadustat, is known to play roles beyond erythropoiesis. Preclinical and some clinical evidence suggests HIF signaling influences bone metabolism (potentially affecting osteoblast differentiation and mineralization) and neurological function (possibly through pathways like CREB/BDNF involved in memory and mood regulation). However, the specific clinical effects of Roxadustat on bone health (density and turnover markers) and neuropsychiatric aspects (depression, anxiety, nerve/muscle structure) in ESKD patients on hemodialysis remain largely unexplored. This study aims to address this gap by evaluating these potential pleiotropic effects of Roxadustat in this patient population.

Study Design and Methods:

This is a randomized, controlled, open-label clinical trial conducted at the Urology and Nephrology Center, Mansoura University, Egypt. Forty-six eligible ESKD patients maintained on chronic hemodialysis for over 3 months will be recruited after providing informed consent.

Patients will be randomized 1:1 into two groups:

Intervention Group (n=23): Patients will receive oral Roxadustat (Evernzo) according to prescribing guidelines, in addition to their standard care (excluding other ESAs).

Control Group (n=23): Patients will continue receiving conventional anemia management (likely including ESAs and/or iron as per standard practice) and standard care.

The follow-up duration for each patient will be 6 months.

Assessments:

All participants will undergo baseline assessments and follow-up evaluations.

Clinical: Full medical history, clinical examination including Handgrip test.

Laboratory: Monthly measurements of serum creatinine, BUN, calcium, phosphorus, magnesium, random blood sugar, venous blood gases, alkaline phosphatase, and albumin. Intact parathyroid hormone (iPTH) and 25-hydroxy vitamin D levels will be measured every 3 months. Fibroblast growth factor 23 (FGF-23) will be measured at baseline and at the end of the study (6 months). Hemoglobin levels will be monitored regularly to guide anemia management.

Radiological: Quantitative computed tomography (QCT) of the lumbar spine will be performed at baseline and 6 months to assess cortical and trabecular bone mineral density (BMD) and volume. A solid phantom composed of calcium hydroxyapatite will be used for calibration.

Psychiatric: Patients will complete the Hamilton Depression Rating Scale (HDRS) and Hamilton Anxiety Rating Scale (HARS) at baseline, 3 months, and 6 months.

Neuromuscular: Musculoskeletal ultrasound (MSK-US) will be performed at baseline and 6 months to evaluate peripheral nerves (diameter, echogenicity, vascularity, morphology) and muscles (architecture, atrophy, echogenicity).

Analysis:

Data will be analyzed using appropriate statistical methods (including t-tests, Mann-Whitney U test, Chi-square/Fisher's exact tests) to compare changes in bone parameters (QCT, bone turnover markers), psychiatric scores (HDRS, HARS), and neuromuscular ultrasound findings between the Roxadustat group and the control group over the 6-month study period. A p-value ≤0.05 will be considered statistically significant. SPSS version 24 will be used for analysis.

This study will provide valuable insights into the broader effects of Roxadustat beyond erythropoiesis, potentially impacting the management of bone and neuropsychiatric complications in hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* The age of the patient is more than 18.
* Patients who are willing to sign informed consent.
* Patients with ESKD on chronic hemodialysis for more than 3 months.

Exclusion Criteria:

* Current pregnancy or lactation.
* Patients with pre-existing malignancy.
* patients with psychosis.
* Known history of hematological disorders or other causes of anemia other than CKD.
* Taking medications that may significantly affect or interact with bone metabolism such as osteo-anabolics or bone resorptives during the last 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in Lumbar Spine Bone Mineral Density | Baseline and 6 months
  Change from baseline in cortical and trabecular bone mineral density (BMD) and volume assessed at the lumbar spine using Quantitative Computed Tomography (QCT). Measured typically in mg/cm³.

SECONDARY OUTCOMES:
Change in Peripheral Nerve Morphology via Ultrasound | Baseline and 6 months
  Change from baseline in cross-sectional area of selected peripheral nerves assessed using Musculoskeletal Ultrasound (MSK-US).
Change in Muscle Morphology via Ultrasound | Baseline and 6 months
  Change from baseline in selected muscles echogenicity assessed using Musculoskeletal Ultrasound (MSK-US).
Change in Handgrip Strength | Baseline and 6 months
  Change from baseline in muscle function as measured by Handgrip Strength test (e.g., measured in kilograms).

CONTACTS AND LOCATIONS:
Locations (1):
- Urology and Nephrology Center, Mansoura University, Al Mansurah, Dakahliya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
A final decision regarding the sharing of individual participant data (IPD) has not yet been made. Factors such as institutional policies, data privacy regulations, resource availability for data de-identification and sharing, and specific requests from qualified researchers will be considered post-study completion before determining if and how IPD might be shared. Any potential sharing would be subject to appropriate ethical and institutional approvals

REFERENCES:
- [Background] Liu Y, Wang J, Chen D, Kam WR, Sullivan DA. The Role of Hypoxia-Inducible Factor 1alpha in the Regulation of Human Meibomian Gland Epithelial Cells. Invest Ophthalmol Vis Sci. 2020 Mar 9;61(3):1. doi: 10.1167/iovs.61.3.1. PMID 32150252
- [Background] Sanghani NS, Haase VH. Hypoxia-Inducible Factor Activators in Renal Anemia: Current Clinical Experience. Adv Chronic Kidney Dis. 2019 Jul;26(4):253-266. doi: 10.1053/j.ackd.2019.04.004. PMID 31477256
- [Background] Zhou Q, Mao M, Li J, Deng F. The efficacy and safety of roxadustat for anemia in patients with dialysis-dependent chronic kidney disease: a systematic review and meta-analysis. Ren Fail. 2023 Dec;45(1):2195011. doi: 10.1080/0886022X.2023.2195011. PMID 37489561